CLINICAL TRIAL: NCT00244959
Title: Surrogate Markers of Response: A Phase II Study of Changes in Breast Density Among Postmenopausal Women Receiving Adjuvant Anastrozole Therapy
Brief Title: Anastrozole in Treating Postmenopausal Women With DCIS or Stage I-III Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0365 CDR0000446285; P30CA006973 (NIH); JHOC-J0365 (Other: SKCCC at Johns Hopkins); JHOC-SKCCC-J0365 (Other: SKCCC at Johns Hopkins)
Record Dates: First submitted 2005-10-25; First posted 2005-10-27 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; ductal breast carcinoma in situ; breast cancer in situ
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — Anastrozole; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anastrozole (Experimental): Anastrozole (1mg, orally, daily) for 12 months as adjuvant therapy for breast cancer
  Interventions: Drug: anastrozole; Procedure: adjuvant therapy

INTERVENTIONS:
Drug: anastrozole — 1 mg orally daily for 12 months
  Other Names: Arimidex
Procedure: adjuvant therapy — treatment received after breast cancer surgery

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using anastrozole may fight breast cancer by lowering the amount of estrogen the body makes.

PURPOSE: This phase II trial is studying how anastrozole effects postmenopausal women who have undergone surgery for ductal carcinoma in situ or stage I, stage II, or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 12-month change in breast density in postmenopausal women with ductal carcinoma in situ (DCIS) or stage I-III breast cancer treated with adjuvant anastrozole.

Secondary

* Determine the change in estrone sulfate levels in patients treated with this drug.
* Correlate the change in breast density with the change in circulating estrone sulfate levels in patients treated with this drug.
* Determine the frequency of polymorphisms in aromatase (CYP19) and evaluate the relationship between wild-type aromatase enzyme with change in breast density and change in estrone sulfate levels in patients treated with this drug.
* Determine the 12-month change in bone density, and correlate it with the change in circulating estrone sulfate levels in patients treated with this drug.
* Correlate the reversal of hypermethylation with change in circulating estrone sulfate levels and breast density in patients treated with this drug.

OUTLINE: This is a pilot study. Patients are stratified according to concurrent bisphosphonate use (yes vs no).

Patients receive oral anastrozole once daily for up to 12 months in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer meeting 1 of the following criteria:

  * Ductal carcinoma in situ (DCIS)
  * Invasive carcinoma

    * Stage I-III disease
* Must have undergone breast cancer surgery within the past 6 months, including any of the following:

  * Mastectomy or lumpectomy with or without radiation
  * Sentinel node and/or axillary node dissection
  * Re-excision of lumpectomy margins
* Intact contralateral breast

  * No prior radiation therapy or mastectomy
  * Prior biopsies allowed
* Hormone receptor status:

  * Estrogen and/or progesterone receptor-positive tumor by immunohistochemical staining

PATIENT CHARACTERISTICS:

Sex

* Female

Menopausal status

* Postmenopausal, defined as 1 of the following:

  * At least 60 years of age
  * Less than 60 years of age and amenorrheic ≥ 12 months prior to study entry
  * Less than 60 years of age, amenorrheic for < 12 months prior to day 1, and luteinizing hormone (LH) and follicle stimulating hormone (FSH) values within postmenopausal range
  * Less than 60 years of age, without a uterus, and LH and FSH values within postmenopausal range
  * Underwent prior bilateral oophorectomy
  * Underwent prior radiation castration AND amenorrheic for ≥ 6 months

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

PRIOR CONCURRENT THERAPY:

Chemotherapy

* No prior or concurrent adjuvant chemotherapy for breast cancer

Endocrine therapy

* No prior aromatase inhibitor
* At least 6 weeks since prior and no concurrent tamoxifen
* At least 6 weeks since prior and no concurrent hormone replacement therapy

  * Concurrent low-dose, local vaginal estrogen in the form of either a conjugated estrogen ring or other similar product (e.g., Estring® or Vagifem®) allowed
* At least 6 weeks since prior and no other concurrent selective estrogen receptor modulators (e.g., raloxifene)

Radiotherapy

* See Disease Characteristics

Surgery

* See Disease Characteristics
* No contralateral breast implant

Other

* Concurrent bisphosphonates allowed at the discretion of the treating oncologist
* No concurrent consumption of soy supplements

  * Concurrent routine dietary consumption of soy-containing foods allowed
* No other concurrent investigational or commercial drugs or therapies for the treatment of DCIS or invasive breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2004-01; Primary Completion 2007-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Change in breast density after 12 months of treatment | 12 months

SECONDARY OUTCOMES:
Change in hormone levels after 12 months of treatment | 12 months
Comparison between change in breast density with change in hormone levels after 12 months of treatment | 12 months
Comparison between the frequency of aromatase polymorphisms with changes in breast density and hormone levels after 12 months of treatment | 12 months
Comparison between change in bone density with change in hormone levels after 12 months of treatment | 12 months
Comparison between tissue methylation with changes in breast density and hormone levels after 12 months of treatment | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Vered Stearns, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Result] Prowell TM, Blackford AL, Byrne C, Khouri NF, Dowsett M, Folkerd E, Tarpinian KS, Powers PP, Wright LA, Donehower MG, Jeter SC, Armstrong DK, Emens LA, Fetting JH, Wolff AC, Garrett-Mayer E, Skaar TC, Davidson NE, Stearns V. Changes in breast density and circulating estrogens in postmenopausal women receiving adjuvant anastrozole. Cancer Prev Res (Phila). 2011 Dec;4(12):1993-2001. doi: 10.1158/1940-6207.CAPR-11-0154. Epub 2011 Sep 1. PMID 21885816